CLINICAL TRIAL: NCT00667628
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of TAC-101 in Combination With Transcatheter Arterial Chemoembolization (TACE) Versus TACE Alone in Japanese Patients With Advanced Hepatocellular Carcinoma
Brief Title: Phase 2 Study of TAC-101 Combined With Transcatheter Arterial Chemoembolization (TACE) Versus TACE Alone in Japanese Patients With Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to safety concerns.
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAC101-203
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2022-04-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — TAC 101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants were administered with placebo tablets matching to TAC-101 orally, every day on the first 14 days (Days 1 to 14) followed by a 7-day (Days 15 to 21) treatment recovery period. Repeated every 21 days cycle up to new lesions were observed or the participant met a treatment discontinuation criterion.
  Interventions: Drug: Placebo
- TAC-101 (Experimental): Participants were administered with TAC-101 tablets, 20 milligram per day (mg/day) orally for every day on the first 14 days (Days 1 to 14) followed by a 7-day (Days 15 to 21) recovery period (21-day Cycle). Repeated every 21 days cycle up to new lesions were observed or the participant met a treatment discontinuation criterion.
  Interventions: Drug: TAC-101

INTERVENTIONS:
Drug: TAC-101 — Participants received TAC-101 20 mg (2 x 10-mg formulated tablets) administered orally every day with approximately 8 oz. water within 1 hour following a morning meal for 14 days followed by a 7-day recovery period, repeated every 21 days.
  Arms: TAC-101
Drug: Placebo — Participants received placebo (two matching tablets) at same frequency and duration of active treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether TAC-101 combined with Transcatheter Arterial Chemoembolization (TACE) is more effective than TACE alone in slowing tumor activity in patients with advanced hepatocellular carcinoma. The study is also looking at the safety of TAC-101 in combination with TACE.

DETAILED DESCRIPTION:
Advanced metastatic hepatocellular carcinoma (HCC) is not treatable by surgical approaches or locoregional therapies such as hepatic artery hemoembolization or radiofrequency ablation (RFA) which are effective in controlling localized tumors. Transcatheter arterial chemoembolization (TACE) is the most commonly performed procedure in the treatment of unresectable liver tumors for selected patients. The TACE procedure delivers highly concentrated drugs to the tumor itself and arrests blood flow. Most patients will have intrahepatic recurrence of their tumors following TACE. Studies of TAC-101, a synthetic retinoid, indicate that although TAC-101 may not induce tumor regression, it appears to have a stabilizing effect, prolonging survival over what was expected historically. This study is designed as a randomized, double-blind, placebo-controlled, parallel-group, phase 2 study in patients with advanced HCC who have undergone a TACE procedure, which will be conducted at multiple sites in Japan, to determine if administration of TAC-101 will enhance the benefits of the TACE procedure.

ELIGIBILITY:
Inclusion Criteria:

- A patient must meet all of the following inclusion criteria to be eligible for enrollment in this study and before undergoing the first TACE procedure of this study:

1. Has an HCC diagnosis by histology or by the following non-invasive criteria observed either at enrollment or in the past.

   * One imaging technique (CT scan or magnetic resonance imaging [MRI] both with unenhanced plus hepatic arterial phase and portal venous phases) showing characteristic features in a focal lesion > 20 mm with arterial vascularization.
   * Two dynamic imaging techniques (CT scan, MRI with unenhanced plus hepatic arterial phase and portal venous phases) showing characteristic features coincidentally in a focal lesion 10-20 mm with arterial vascularization.
2. Is TACE naïve or has received the most recent TACE procedure at least 120 days before signing ICF.
3. Eligible to receive TACE and being scheduled to receive TACE.
4. Must be ≥ 20 years of age.
5. Is not amenable to treatment with curative surgery, transplant, or percutaneous ablation, including RFA, percutaneous ethanol injection therapy (PEIT) and percutaneous microwave coagulation therapy (PMCT).
6. Must have lesions in the liver that are confirmed nodular type with demonstrated substantial hypervascularity by CT scan or MRI both with unenhanced plus hepatic arterial phase and portal venous phases performed prior to first TACE in this study with the following tumor features:

   * If there are ≥ 4 intrahepatic lesions, all lesions can be < 30 mm. or, regardless of the number of lesions, the longest diameter of at least one intrahepatic lesion is ≥ 30 mm).
   * No vascular invasion in main trunk and first order branch of portal vein.
   * No extrahepatic tumor spread. The absence of extrahepatic abdominal tumors must be confirmed.
7. Has adequate organ function as defined by the following criteria: White blood cell (WBC) count > 3,000/mm3; Platelet count > 60,000/mm3; Hemoglobin > 8.0 grams (g)/deciliter (dL); Aspartate transaminase (AST) < 5 x upper limit of normal (ULN); Alanine transaminase (ALT) < 5 x ULN; Total bilirubin < 2.0 mg/dL; Albumin ≥ 2.8 g/dL; Serum creatinine ≤ 1.5 mg/dL; International normalized ratio (INR) ≤ 2.0; Triglyceride ≤ 2.5 x ULN.
8. Must have a Child-Pugh classification of ≤ 8.
9. Must have a Cancer of the Liver Italian Program (CLIP)60 score of 0, 1, 2 or 3 (Appendix B).
10. Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
11. Must be willing and able to comply with schedule visits, treatment plans, laboratory tests, and other study procedures.
12. Must provide written informed consent prior to the implementation of any study assessment or procedures.

Exclusion Criteria:

* Patients will be excluded from participation in the study if any of the following conditions are observed before undergoing the first TACE procedure:

  1. Patient has longest diameter of intrahepatic lesion ≥ 100 mm.
  2. Patient has only infiltration type of HCC.
  3. Patient has extrahepatic metastasis of HCC including regional lymph node metastases (including in lymph nodes and organs).
  4. Patient had systemic chemotherapy (eg, sorafenib, doxorubicin), immunotherapy, or biologic therapy or radiotherapy for HCC, or treatment with TAC-101.
  5. Patient received treatment with any of the following within the specified time frame: Any major surgical procedure within 28 days prior to signing the ICF; Any transfusion, treatment with blood component preparation, albumin preparation, and granulocyte colony stimulating factor (G-CSF) within 14 days prior to signing the ICF; Any local therapy such as alcohol injection, radiofrequency/ultrasound ablation, intraarterial chemotherapy (transcatheter arterial injection) for HCC performed within 28 days prior to signing the ICF; Any investigational agent within 28 days prior to signing the ICF.
  6. Patient has ascites, pleural effusions or pericardial fluid refractory to diuretic therapy.
  7. Patient has clinical symptoms of hepatic encephalopathy.
  8. Patient has active or uncontrolled clinically serious infection excluding chronic hepatitis.
  9. Patient has a history of gastrointestinal (GI) bleeding in last 3 months.
  10. Patient has previous or concurrent malignancy except for in situ carcinoma of the cervix, or other solid tumor treated curatively and without evidence of recurrence for at least 3 years prior to the study.
  11. Patient has uncontrolled metabolic disorders or other nonmalignant organ or systemic diseases or secondary effects of cancer that induce a high medical risk and/or make assessment of survival uncertain.
  12. Patient has any history of deep vein thrombosis (DVT), pulmonary embolism (PE), myocardial infarction (MI), cerebrovascular accident (CVA), transient ischemic attack (TIA), unstable angina pectoris, or any other significant thromboembolic event (TE) during the last 3 years.
  13. Patient has clinically significant electrocardiogram (ECG) abnormality.
  14. Patient has GI disease resulting in an inability to take oral medication.
  15. Patient has known allergy or hypersensitivity to TAC-101, doxorubicin, epirubicin, other anthracyclines, anthracenediones or any of the components used in the study drug formulations.
  16. Patient has known hypersensitivity to iodinated contrast medium.
  17. Patient is receiving therapeutic regimens of anticoagulants. However, use of low dose anticoagulants for prophylactic care of indwelling venous access device is permitted.
  18. Patient is taking medication known or suspected to predispose patient to an increased risk of VTE (eg, oral contraceptives, hormone replacement therapy, megestrol acetate).
  19. Patient is taking azoles or tetracyclines, because of the potential for drug interactions.
  20. Women who intend to become pregnant or are pregnant or lactating and men able to procreate that refuse to use a highly effective method of birth control during treatment with study medication and up to 6 months thereafter.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-04-24 (Actual); Primary Completion 2009-12-22 (Actual); Study Completion 2009-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Central, MD, Study Director — Taiho Oncology, Inc.
Locations (29):
- Japan (29):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National hospital organization Shikoku Cancer Center, Matsuyama, Ehime
  - Fukuoka University Hospital, Jonan-ku, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Ogaki Municipal Hospital, Oogaki, Gifu
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - Asahikawa-Kosei General Hospital, Asahikawa, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - The Hospital of Hyogo College of Medicine, Hishinomiya, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital, Morioka, Iwate
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Nara Medical University Hospital, Kashihara, Nara
  - Okayama University Hospital, Shikata-cho, Okayama-ken
  - Osaka City University Hospital, Abeno-ku, Osaka
  - Osaka medical Center for Cancer and Cardiovascular Diseases, Higashinari-ku, Osaka
  - Osaka City General Hospital, Miyakojima-ku, Osaka
  - Kansai Medical Univesity Takii Hospital, Moriguchi, Osaka
  - Kinki University Hospital, Ōsaka-sayama, Osaka
  - Osaka Red Cross Hospital, Tennoji-ku, Osaka
  - Shizuoka Cancer Center Hospital, Sunto-gun, Shizuoka
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Kyoundo Hospital, Chiyoda City, Tokyo
  - Tochigi Cancer Center, Chiyoda-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Wakayama Medical University Hospital, Kimiidera, Wakayama
  - Kochi Health Science Center, Kochi
  - Kumamoto University Hospital, Kumamoto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 67 participants were screened, of which 54 participants received the first transcatheter arterial chemoembolization (TACE) prior to randomization. Two participants discontinued prior to randomization due to adverse event and thus, a total of 52 participants were randomized in the study and received study drug in the double-blind period. The study was prematurely terminated by the Sponsor due to safety concerns.
Pre-assignment Details: Randomization was balanced between treatment arms according to the stratification factors of number of lesions (less than [<] 5 versus greater than equal to [>=] 5) and baseline alpha-fetoprotein (AFP) level (<400 nanograms per milliliters [ng/mL] versus >=400 ng/mL).
Groups:
- Placebo: Participants were administered with placebo tablets matching to TAC-101 orally, every day on the first 14 days (Days 1 to 14) followed by a 7-day (Days 15 to 21) treatment recovery period (21-day Cycle). Repeated every 21 days up to new lesions were observed or the participant met a treatment discontinuation criterion.
- TAC-101: Participants were administered with TAC-101 tablets, 20 milligrams per day (mg/day) orally for every day on the first 14 days (Days 1 to 14) followed by a 7-day (Days 15 to 21) recovery period (21-day Cycle). Repeated every 21 days up to new lesions were observed or the participant met a treatment discontinuation criterion.
Period: Overall Study
Arm/Group | Placebo | TAC-101
Started | 25 | 27
Completed | 0 | 0
Not Completed | 25 | 27
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 6 | 6
Not completed — Investigator Considers in Best Interest | 1 | 0
Not completed — Sponsor Terminated Study | 17 | 21

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who underwent a first combination with transcatheter arterial chemoembolization (TACE) procedure prior to randomization in this study, who were randomized and received at least one dose of double-blind medication.
Groups:
- TAC-101: Participants were administered with TAC-101 tablets, 20 mg/day orally for every day on the first 14 days (Days 1 to 14) followed by a 7-day (Days 15 to 21) recovery period (21-day Cycle). Repeated every 21 days cycle up to new lesions were observed or the participant met a treatment discontinuation criterion.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAC-101 | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.77) | 69.4 (8.31) | 69.1 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 22 | 23 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 27 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Appearance of New Lesions (TTNL)
Description: TTNL was defined as the time from the date of randomization to the date of appearance of a new lesion. Participants who had no appearance of new lesions had their TTNL censored at the date of their last tumor assessment.
Time Frame: From randomization (within 14 days prior to first TACE) assessed every 9 weeks after first TACE to date of appearance of a new lesion or until cut-off date (22-Dec-2009) (up to approximately 20 months)
Population: Safety population included all participants who underwent a first combination with TACE procedure prior to randomization in this study, who were randomized and who received at least one dose of double-blind medication. Here, overall number of participants analyzed' signifies participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: months
Groups:
- TAC-101: Participants were administered with TAC-101 tablets, 20 mg/day orally for every day on the first 14 days (Days 1 to 14) followed by a 7-day (Days 15 to 21) recovery period (21-day Cycle). Repeated every 21 days up to new lesions were observed or the participant met a treatment discontinuation criterion.
Arm/Group | Placebo | TAC-101
Number analyzed (Participants) | 24 | 26
months | 8.4 (4.00) | 7.0 (4.07)

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to date of death. Participants who were still alive at the time of analysis had their survival time censored at the last date known to be alive.
Time Frame: From randomization (within 14 days prior to first TACE) assessed every 9 weeks after first TACE until cut-off date of 22 Dec 2009 (up to approximately 20 months)
Population: Safety population included all participants who underwent a first combination with TACE procedure prior to randomization in this study, who were randomized and who received at least one dose of double-blind medication.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | TAC-101
Number analyzed (Participants) | 25 | 27
months | 13.9 (2.87) | 13.2 (4.18)

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from date of randomization to the date of disease progression (radiological, only).
Time Frame: as for outcome 2
Population: The safety population was planned, with an independent review of tumor response. However, the independent reviews were deferred. Hence, the data was not collected and not evaluated.
Arm/Group | Placebo | TAC-101
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Objective Tumor Response Rate (ORR)
Description: ORR was defined as the percentage of participants with objective evidence of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than (<)10 millimeters (mm). PR was defined as at least a 30 percent decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters.
Time Frame: as for outcome 2
Population: The safety population was planned, with an independent review of tumor response. However, the independent reviews were deferred. Hence, the data were not collected and not evaluated.
Arm/Group | Placebo | TAC-101
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Plasma Levels of Tumor Marker Alpha-fetoprotein (AFP)
Description: AFP was known as a tumor marker for advanced hepatocellular carcinoma (HCC) and was recognized as useful for following the course of HCC. Changes in serum AFP parallel the clinical course of HCC, where elevations can precede clinical deterioration and tumor recurrence.
Time Frame: Baseline, End of treatment (last dose of study medication, i.e., approximately 7 months)
Population: Safety population included all participants who underwent a first combination with TACE procedure prior to randomization in this study, who were randomized and who received at least one dose of double-blind drug. Here, 'overall number of participants analyzed' signifies participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Placebo | TAC-101
Number analyzed (Participants) | 24 | 24
nanogram per milliliter (ng/mL) | -324.0 (1903.05) | 8147.9 (37555.15)

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: Any untoward medical condition that occurs in a participants while participating in a clinical study and does not necessarily have a causal relationship with the use of the study drug was considered an adverse event (AE). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs: AEs that occur from the initiation of any study treatment administration, and do not necessarily have a causal relationship to the use of the study drug.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug or until the start of new anti-tumor therapy, whichever was earlier (up to approximately 8.5 months)
Population: Safety population included all participants who had underwent a first combination with TACE procedure prior to randomization in this study, who were randomized and who had received at least one dose of double-blind medication.
Measure: Number; unit: participants
Arm/Group | Placebo | TAC-101
Number analyzed (Participants) | 25 | 27
participants
  TEAEs | 22 | 25
  TESAEs | 2 | 5

ADVERSE EVENTS:
Time Frame: AEs were collected from first dose (i.e., Day 1) of study drug to last dose of study drug + 30 days (up to approximately 8.5 months). Deaths were collected from Baseline up to end of study (up to approximately 20 months).
Description: Reported AEs were TEAEs that developed/worsened in grade or became serious during TEAE period (defined as the time from the first dose of study drug to the last dose of study drug + 30 days) and was assessed on safety population. All-Cause Mortality data collected during the study was assessed for all randomized participants.
Arm/Group | Placebo | TAC-101
All-Cause Mortality (participants affected / at risk) | 6/25 | 6/27
Serious Adverse Events (participants affected / at risk) | 2/25 | 5/27
Other Adverse Events (participants affected / at risk) | 22/25 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | TAC-101 (N=27)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Contralateral breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | TAC-101 (N=27)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 6 (9) | 7 (10)
Oedema peripheral (General disorders) | 2 (3) | 1 (1)
Pyrexia (General disorders) | 6 (8) | 5 (8)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 2 (2)
Fibrin d dimer increased (Investigations) | 1 (1) | 3 (3)
Thrombin-antithrombin iii complex increased (Investigations) | 0 (0) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 10 (12)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was terminated early due to the unexpected higher occurrence of thromboembolic events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes